CLINICAL TRIAL: NCT05280392
Title: Expectation, Motivation and Experience of HIV-patients Regarding Participation to the EHVA T02/ANRS VRI 07 HIV Cure-related Clinical Trial (AMEP-EHVA T02)
Brief Title: Expectation, Motivation and Experience of HIV-patients Regarding Participation to an HIV Cure-related Clinical Trial
Acronym: AMEP-EHVA T02
Status: Terminated | Type: Observational
Why Stopped: EHVA T02/ANRS VRI07 clinical trial had been discontinued. Find relevant information on the EHVA website: https://ehv-a.eu/trials/ehva-t02
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: ANRS 95052
Record Dates: First submitted 2022-02-11; First posted 2022-03-15 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: HIV Seropositivity
Keywords: HIV cure-related clinical trials; Participants' expectations and experiences
MeSH Terms: conditions — HIV Seropositivity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- People living with HIV: PLWH who were offered to participate in the EHVA T02/ANRS VRI07 clinical trial
  Interventions: Other: Self-administered questionnaires; Other: Semi-directive individual interviews

INTERVENTIONS:
Other: Self-administered questionnaires — 4 self-questionnaires given to EHVA T02 participants: at inclusion (Q1, week 0), at the beginning of the ATI period (Q2, week 18), at the end of the ATI period (Q3, date depending on the participant) and at the end of the follow-up period of the clinical trial (Q4, week 54 at the latest)
Other: Semi-directive individual interviews — With EHVA T02 participants (n=10 to 15): at the end of the follow-up period of the clinical trial.
Other: Semi-directive individual interviews — With patients who refused to participate to EHVA T02 or patients not included because of negative screening results (n=10 to 15): within 21 days after the refusal or the results of the screening

SUMMARY:
Following the ANRS-APSEC survey, AMEP-EHVA T02 is a longitudinal social science study that will explore the experience of people living with HIV (PLWH) who were offered to participate in the European randomized phase II placebo-controlled trial of vedolizumab with or without therapeutic HIV MVA vaccine including antiretroviral treatment interruption (EHVA T02/ANRS VRI07).

DETAILED DESCRIPTION:
Moving towards the discovery of an HIV cure is of major public health interest, not only for people living with HIV (PLWH) who currently must take lifelong antiretroviral treatment (ART), with its associated side effects and comorbidities, but also for the community as a whole. An HIV cure will end the virus transmission, lead to global care-related savings and decrease in HIV-related stigma.

The present longitudinal social science study concerns the experience of PLWH who were offered to participate in the European randomized phase II placebo-controlled trial of vedolizumab with or without therapeutic HIV MVA vaccine including ART treatment interruption (EHVA T02/ANRS VRI07).

The objectives are to document:

1. the evolution over time of expectations and motivations related to participation in the trial,
2. anticipation and understanding of risks and benefits related to participation,
3. evolution over time of participation experience and of satisfaction with the information delivered,
4. experience and perception of the ATI period and its impact on preventive behaviours and sexual quality of life,
5. motivations and experience related to refusal of participation, or if any, related to non-inclusion because of negative screening results.

This international multicentre longitudinal study will be nested within the EHVA T02/ANRS VRI07 trial, and will comprise two components. A quantitative component designed to answer to the four first objectives, and a qualitative one that will retrospectively deepen the trial participation experience and will also document the motivation for participation refusal and the experience of participants not included because of negative screening results (objective 5). The quantitative survey will be conducted within participating centres that estimate to include at least 5 participants, and the qualitative one only in France for feasibility purpose.

ELIGIBILITY:
Inclusion Criteria:

* people living with HIV
* who were offered to participate in EHVA T02 clinical trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The quantitative survey will be proposed to all the PLWH included in the EHVA T02/ANRS VRI07 trial (except in germany where the center estimates to include less than 5 participants)(n = 69 max), the inclusion criteria being those defined by the clinical protocol.
  Participants to the qualitative survey will be recruted in the three EHVA T02/ANRS VRI07 French centers.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2022-06-21 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Proportion of patients satisfied with their participation and the associated factors | through study completion, an average of 1 year
  Through statistical analyses of some self-administered questionnaires items we will highlight the participants' satisfaction and experience of the participation.
Impact of the participation in the trial on participant quality of life and quality of sexual life | through study completion, an average of 1 year
  Through statistical analyses of some self-administered questionnaires items (in particular the SF12.v2 scale for quality of life) and thematic analyses of semi-directive individual interviews we will highlight the impact of the participation in the trial.

CONTACTS AND LOCATIONS:
Overall Officials: Christel Protiere, Dr, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, UMR1252 SESSTIM, France
Locations (1):
- CHUV, Lausanne, Switzerland